CLINICAL TRIAL: NCT01856894
Title: Is Serum Anti-Mullerian Hormone (AMH) Level Associated With Body Weight, Glycemic and Lipidemic Markers in Adolescent Girls With Polycystic Ovaries?
Brief Title: Serum Anti-Mullerian Hormone (AMH) Levels in Overweight and Obese Adolescent Girls With Polycystic Ovaries
Status: Completed | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: PCODHC
Record Dates: First submitted 2013-05-14; First posted 2013-05-20 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Polycystic Ovary Syndrome
Keywords: polycystic ovary syndrome; Anti-Mullerian Hormone; obesity
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In this study the investigators aimed to investigate whether there is a relation between body weight and serum anti mullerian hormone levels in adults with polycystic ovary syndrome. For this purpose the investigators designed a prospective study including three groups. The group I is defined as adults with polycystic ovary syndrome and body mass index is greater than 25. The group II is defined as adults with polycystic ovary syndrome and body mass index is less than 25. The group III is defined as adults with non-polycystic ovary syndrome and body mass index is less than 25. The all three groups are compared considering their serum AMH levels,lipid profiles, sex steroids and glycemic analyses.

DETAILED DESCRIPTION:
In this study the investigators aimed to investigate whether there is a relation between body weight and serum anti mullerian hormone levels in adults with polycystic ovary syndrome. For this purpose the investigators designed a prospective study including three groups. The diagnosis of polycystic ovary syndrome was made in the presence of ;oligo- and/or anovulation,clinical and/or biochemical signs of hyperandrogenism and polycystic ovaries. Clinical hyperandrogenism was defined by the presence of hirsutism , acne, or the presence of androgenic alopecia , biochemical hyperandrogenemia was defined as a serum level of total testosterone higher than 2.60 nmol/L, body mass index (BMI) was calculated as weight in kilograms divided by the square of height in meters. The patients were classified as obese with BMI ≥ 25 kg/m2 , adolescent patients were diagnosed 2 years after menarche in order to avoid the misdiagnosis of transitory functional hyperandrogenism and menstrual disorders during puberty. The all three groups are compared considering their serum AMH levels,lipid profiles, sex steroids and glycemic analyses.

ELIGIBILITY:
Inclusion Criteria:

The participants with the following findings;oligo- and/or anovulation, clinical and/or biochemical signs of hyperandrogenism and polycystic ovaries, presence in each ovary of 12 or more follicles measuring 2-9 mm in diameter and/or increased ovarian volume (> 10 mL).

Exclusion Criteria:

The participants with the following findings;pregnancy,breastfeeding,known liver disease or alanine aminotransferase (60 IU/l), creatinine (130 mmol/l), known alcohol abuse, diabetes mellitus and treatment with oral glucocorticoids or hormonal contraceptives.

Patients could be included if hormonal contraception had been discontinued at least 1 month previously.

Ages: 12 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The diagnosis of Polycystic ovary syndrome was made in the presence of ;oligo- and/or anovulation,clinical and/or biochemical signs of hyperandrogenism and polycystic ovaries. Clinical hyperandrogenism was defined by the presence of hirsutism, acne, or the presence of androgenic alopecia , biochemical hyperandrogenemia was defined as a serum level of total testosterone higher than 2.60 nmol/L, body mass index (BMI) was calculated as weight in kilograms divided by the square of height in meters. The patients were classified as obese with BMI ≥ 25 kg/m2 , adolescent patients were diagnosed 2 years after menarche in order to avoid the misdiagnosis of transitory functional hyperandrogenism and menstrual disorders during puberty.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2013-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Ovarian reserve, as measured by basal follicle stimulating hormone/anti-Mullerian hormone/antral follicle count | Three months

SECONDARY OUTCOMES:
Body weight | Three months

CONTACTS AND LOCATIONS:
Overall Officials: Hüseyin Cengiz, M.D., Study Director — Bakirkoy Dr Sadi Konuk Teaching and Research Hospital, Department of Obstetrics and Gynecology; Cihan Kaya, M.D., Principal Investigator — Bakirkoy Dr Sadi Konuk Teaching and Research Hospital, Department of Obstetrics and Gynecology; Şükrü Yıldız, M.D., Principal Investigator — Bakirkoy Dr Sadi Konuk Teaching and Research Hospital, Department of Obstetrics and Gynecology; Hediye Dağdeviren, M.D., Principal Investigator — Bakirkoy Dr Sadi Konuk Teaching and Research Hospital, Department of Obstetrics and Gynecology
Locations (1):
- Bakirkoy Dr Sadi Konuk Teaching and Research Hospital, Department of Obstetrics and Gynecology, Istanbul, Turkey (Türkiye)